[Unique Protocol ID: Dh3108103/64] (October 5, 2021)
Official Title: Clinical Results of Minimally Invasive Plate Osteosynthesis Versus Conventional Approach in Volar
Locking Plate for Close Fractures of Distal End Radius Under WALANT

| Code |
|------|
| Coue |

(Witness: .....)

## **Informed Consent Form**

| Informed Consent Form |
|---|
| Clinical Results of Minimally Invasive Plate Osteosynthesis versus Conventional Approach in Volar Locking Plate for Close Fractures of Distal End Radius under WALANT |
| Date of Signing: |
| - Before signing this consent form, I have been explained by the researcher about the purpose of the research, research methods, potential risks or side effects from the research or medications used, as well as the expected benefits in detail. I understand these thoroughly. |
| - The researcher assures that they will willingly answer any questions I may have and will not withhold information until I am satisfied. |
| - I voluntarily participate in this research without coercion or inducement. |
| - I have the right to withdraw from the study at any time, and this withdrawal will not affect the medical treatment I am currently receiving or will receive in the future. |
| - The researcher assures that information about me will be kept confidential and will only be disclosed in the form of research summaries without revealing my name. Disclosure of information to relevant organizations will only be done for academic reasons. |
| - In the event of any harm resulting from the research, I will receive medical treatment as specified in the information provided to research participants. |
| - I will receive one set of informational documents related to the research. |
| - I acknowledge and understand the above statements and willingly sign this consent form. |
| Signature: (Name in block letters:) |
| Signature: (Name of Researcher: Mr. Suphasan Keatisuwan) |
| Signature: (Witness:) |
| Signature: |